CLINICAL TRIAL: NCT00286572
Title: Comparison in Survival in Patients With Insulin-dependent and Non-insulin-dependent Diabetes Mellitus With Known or Suspected Coronary Artery Disease Undergoing Major Non-cardiac Surgery
Brief Title: Long-term Mortality in Diabetics Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Daniel Bolliger, PD Dr. Daniel Bolliger, University Hospital, Basel, Switzerland
Other Study IDs: 129/03
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus; Coronary Heart Disease; Major Non-cardiac Surgery
Keywords: insulin-dependent diabetes mellitus; non-insulin-dependent diabetes mellitus; coronary artery disease; long-term mortality
MeSH Terms: conditions — Diabetes Mellitus; Coronary Disease; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with CAD and diabetes mellitus have a better prognosis than patients with CAD and no diabetes mellitus. In acute coronary syndrome patients with an insulin therapy had a better survival than patients with oral antidiabetics. But there is not known wether perioperative therapy with insulin or oral antidiabetics is associated with higher risk for higher perioperative cardiac morbidity and mortality and worse long-term survival.

DETAILED DESCRIPTION:
Diabetes mellitus is an important risk factor for arteriosclerosis in general and for coronary artery disease. Patients with CAD have a worse prognosis if they have diabetes mellitus. But it is not known whether the treatment of Dm has an influence on mortality or morbidity.

In face of the high number of patients with Dm and the therapeutic consequences this prospective study wants to compare short-time and long-time morbidity in Patients with Dm undergoing major non-vascular surgery. Inclusion criteria are medically treated Dm (insulin or oral antidiabetics) and major non cardiac surgery.

The "normal" perioperative treatment of the study is not changed by the study itself.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus with insulin or oral antidiabetics
* proven coronary artery disease or very high risk for it
* major non-vascular surgery

Exclusion Criteria:

* emergency
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treated diabetes mellitus undergoing surgery with major risk or patients with treated diabetes mellitus and known coronary artery disease undergoing surgery with major or intermediate risk
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2004-01; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Death and/or major adverse cardiac events | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Filipovic, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, CH, Switzerland